CLINICAL TRIAL: NCT07283406
Title: Effect of High-intensity Interval Training on Cardiometabolic Health and Physical Fitness in Young Adults With Obesity
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitario de Tlajomulco, Universidad de Guadalajara (Other)
Responsible Party: Principal Investigator, José Manuel Pérez Casillas, Principal Investigator, Centro Universitario de Tlajomulco, Universidad de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUTLAJO251028
Record Dates: First submitted 2025-11-13; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Obesity & Overweight
Keywords: obesity; HIIT; MICT
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT Group (Experimental): This group will train for 12 weeks
  Interventions: Other: High-intensity interval training intervention; Other: Educational sessions
- MICT Group (Active Comparator): This group will train for 12 weeks
  Interventions: Other: Moderate-intensity continuous training intervention; Other: Educational sessions

INTERVENTIONS:
Other: High-intensity interval training intervention — The HIIT group will undergo training for 12 weeks, with a frequency of three sessions per week, completing a total of 36 sessions. Each session will include a 5-minute warm-up and a 5-minute cool-down at 50-60% of maximum heart rate (HRmax). The training protocol will consist of 2-minute high-intensity intervals performed at 90-95% HRmax, corresponding to a Borg rating of perceived exertion (RPE) of 17-18, alternated with 2-minute recovery periods at 70% HRmax (RPE 12-14). A total of five intervals will be completed per session, resulting in an overall high-intensity workload of 18 minutes. All training sessions will be conducted on a stationary cycle ergometer
  Arms: HIIT Group
Other: Moderate-intensity continuous training intervention — The MICT group will perform moderate-intensity continuous training at 60-70% HRmax, corresponding to an RPE of 12-14, for 35-45 minutes on a stationary cycleergometer. Heart rate and physical activity levels will be continuously monitored in both groups using a chest-strap heart rate sensor (Polar H9, Polar Electro, Finland).
  Arms: MICT Group
Other: Educational sessions — In addition, four educational sessions will be conducted to provide dietary recommendations to all participants. These sessions will aim to promote balanced eating habits and to discourage the excessive consumption of ultra-processed foods or alcohol, as these factors could interfere with the intervention outcomes.

SUMMARY:
The objective of the present project is to compare the effects of two types of training on cardiovascular health components and physical fitness in young adults with obesity.

DETAILED DESCRIPTION:
Obesity represents a serious public health problem, and its prevalence continues to rise worldwide. Numerous studies have documented the positive effects of moderate-intensity continuous training (MICT) on cardiovascular and metabolic health in individuals living with obesity; however, the effects of high-intensity interval training (HIIT) are still being explored.

Therefore, the objective of the present research protocol is to analyze and compare the effects of an MICT program and an HIIT program on cardiometabolic biomarkers and physical fitness in young adults with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Young adults
* BMI ≥ 30 kg/m^2" and < 40 kg/m^2
* Signed informed consent form

Exclusion Criteria:

* Participants who smoke
* Clinical diagnosis of hypothyroidism
* Clinical diagnosis of type 1 diabetes mellitus
* Clinical diagnosis of type 2 diabetes mellitus
* Clinical diagnosis of grade 3 obesity
* Clinical diagnosis of hypertension
* Clinical diagnosis of acute myocardial infarction or angina pectoris
* Use of nitrates and calcium channel blockers within 4 days prior to the start of the study
* Use of beta-blockers or hypoglycemic agents within 7 days prior to the intervention
* Pregnant women
* Breastfeeding women
* Men consuming more than 40 g of alcohol per day or women consuming more than 20 g per day
* Postural and biomechanical disorders (knee, foot, and spine)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-03 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Maximum oxygen uptake (VO₂max) | Baseline and after 12 weeks
  VO₂max (ml/min/kg): Change from Baseline at 12 weeks, measured using a submaximal exercise test based on the Åstrand-Ryhming protocol
Weight | Baseline and after 12 weeks
  Weight (kg): Changes in weight from baseline to 12 weeks of intervention.
Height | Baseline and after 12 weeks
  Height (cm): Changes in height from baseline to 12 weeks of intervention.
Body mass index (BMI) | Baseline and after 12 weeks
  BMI (kg/m2): Change from Baseline at 12 weeks, calculated by: weight (kg)/ height (m^2)
Body fat percentage | Baseline and after 12 weeks
  Body fat percentage (%): Changes in body fat assessed by bioelectrical impedance analysis (BIA)
Muscle mass percentage | Baseline and after 12 weeks
  Muscle mass percentage (%): Changes in muscle mass measured using bioelectrical impedance analysis (BIA)
Waist circumference | Baseline and after 12 weeks
  Waist circumference (cm): Changes in waist circumference will be measured using a Lufkin measuring tape (USA) following the guidelines of the International Society for the Advancement of Kinanthropometry (ISAK)
Waist-to-hip ratio | Baseline and after 12 weeks
  Waist-to-hip ratio: Changes in waist-to-hip ratio will be calculated by dividing the waist measurement by the hip measurement
Glucose | Baseline and after 12 weeks
  Glucose (mg/dl): Changes from baseline to 12 weeks of intervention
Triglycerides | Baseline and after 12 weeks
  Triglycerides (mg/dl): Changes from baseline to 12 weeks of intervention
Total cholesterol | Baseline and after 12 weeks
  Total cholesterol (mg/dl): Changes from baseline to 12 weeks of intervention
HDL cholesterol | Baseline and after 12 weeks
  HDL cholesterol (mg/dl): Changes from baseline to 12 weeks of intervention
LDL cholesterol | Baseline and after 12 weeks
  LDL cholesterol (mg/dl): Changes from baseline to 12 weeks of intervention
C-reactive protein (CRP) | Baseline and after 12 weeks
  CRP (mg/dl): Changes from baseline to 12 weeks of intervention
Systolic blood pressure (SBP) | Baseline and after 12 weeks
  SBP (mmHg): Changes from baseline to 12 weeks of intervention
Diastolic blood pressure (DBP) | Baseline and after 12 weeks
  DBP (mmHg): Changes from baseline to 12 weeks of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Universitario de Tlajomulco, Universidad de Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No